CLINICAL TRIAL: NCT05098301
Title: Data Therapy Collection to Evaluate Performances of an Automated Insulin Titration Algorithm Compared to Standard Method of Titration
Acronym: GLUCAL3
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0562
Record Dates: First submitted 2021-10-18; First posted 2021-10-28 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Diabetes
Keywords: Diabetes; Functional insulin therapy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A data collection of blood glucose values, insulin, meal composition will be performed for a period of two months, to evaluate the performances of an automated insulin titration algorithm

ELIGIBILITY:
Inclusion criteria:

* Person with Type 1 diabetes
* Treated by basal-bolus therapy with MDI or pump
* Patient with social security or beneficiary of medical coverage
* Patient using functional insulin therapy or starting and education course
* Patient able to read and understand the procedure, and able to express consent for study protocol

Exclusion criteria:

* Patient abusing substances
* Patient deprived of liberty by judicial or administrative decision, person subject to a legal protection measure, patient having a psychological condition making him unable to follow and understand study protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 1 diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
evaluate the performances of an insulin titration algorithm | day 1
  to evaluate the performances of an insulin titration algorithm to calculate insulin therapy parameters at the same precision of an expert practitioner

SECONDARY OUTCOMES:
measure time-in-range evolution adjustment of insulin therapy parameters | day 1
  to measure time-in-range evolution before and after adjustment of insulin therapy parameters by practitioner

CONTACTS AND LOCATIONS:
Overall Officials: Eric RENARD, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC